CLINICAL TRIAL: NCT00676169
Title: Longitudinal Assessment of Risk Factors For and Impact of Pseudomonas Aeruginosa Acquisition and Early Anti-Pseudomonal Treatment in Children With CF
Brief Title: The EPIC Observational Study
Acronym: EPIC OBS
Status: Completed | Type: Observational
Sponsor: CF Therapeutics Development Network Coordinating Center (Network)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC002
Record Dates: First submitted 2008-05-08; First posted 2008-05-12 (Estimated); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Cystic Fibrosis
Keywords: Pseudomonas aeruginosa; EPIC
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For study purposes, OP swabs or expectorated sputum for bacterial culture will be obtained annually beginning in the calendar year of first isolation of Pa from a respiratory culture at the local site laboratory. A serum sample for serology assessment and banking will be obtained annually in conjunction with a scheduled clinical blood draw whenever possible. Under a separate consent, additional blood (6 ml) will be collected for DNA use and banking for studies of genetic factors that may be associated with CF pathogenesis, disease progression, and clinical outcomes. These studies will test for association between gene variants and various CF-related phenotypes using either a targeted (i.e., candidate gene) approach or by performing a whole-genome scan.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Pa negative or concurrently enrolled in the EPIC Clinical Trial

SUMMARY:
The purpose of this study is to better define risk factors preceding first isolation of Pseudomonas aeruginosa (Pa) from respiratory cultures in cystic fibrosis (CF) lung disease and to better define clinical outcomes associated with acquisition of Pa. This study will also collect and bank DNA samples for current and future studies designed to enhance the understanding of the pathogenesis of CF.

DETAILED DESCRIPTION:
The EPIC Observational Study is a longitudinal, prospective, observational study that was originally conducted at 59 sites. The current five-year extension study is being conducted at 54 sites.

The EPIC Observational Study will serve as a freestanding epidemiologic study of the risk factors for and clinical impact of initial Pa acquisition and anti-pseudomonal therapy. Defining the risk factors for Pa acquisition can potentially allow for preventive measures and identification of high-risk populations requiring closer monitoring. Despite rigorous data collection, previous studies have been limited by small sample sizes and by conduct at one or two centers. This study will include a much larger sample size from many more centers than previous studies. It will thus provide for more generalizable results and more precise risk estimates for previously identified risk factors for Pa acquisition, and it will allow for exploration of novel risk factors not included in earlier studies. Better understanding of the clinical outcomes associated with Pa acquisition and the outcomes associated with different types of anti-pseudomonal therapies will inform the development of rational early intervention treatment regimens. Better knowledge about temporal relationships between respiratory signs and symptoms, Pa serology, and CF airway microbiology may lead to improved strategies for early detection of Pa and could have important implications for the timing of interventions aimed at preventing or treating early Pa acquisition. Finally, this study will serve as an important source of Pa and S. aureus isolates, serum samples, and DNA samples that will be used and banked for studies designed to enhance the understanding of the pathogenesis of CF, e.g., microarray investigations of early Pa isolates, investigations to identify proteomic biomarkers of airway inflammation, and investigations to identify genetic factors related to CF disease progression, including early lung disease, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages less than or equal to 12 years.
* Diagnosis of CF based upon the criteria established by the 1997 CF Consensus Conference: (i) sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis; or (ii) genotype with two identifiable mutations consistent with CF; or (iii) an abnormal nasal transepithelial potential difference, and (iv) one or more clinical features consistent with CF.
* No prior isolation of Pa from respiratory cultures (1 or more cultures in 24 months prior to enrollment), or, if prior isolation of Pa from respiratory cultures, at least a two-year history of Pa negative cultures (1 or more cultures/year), or concurrently enrolled in the EPIC Clinical Trial.
* Signed informed consent to participate in data submission to the CFF National Patient Registry.
* Signed informed consent by parent or legal guardian.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Cystic Fibrosis who are Pa negative or concurrently enrolled in the EPIC Clinical Trial
Sampling Method: Non-Probability Sample
Enrollment: 1248 (Actual)
Dates: Start 2004-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
To better define risk factors for first isolation of Pa from respiratory culture, as well as for emergence of mucoid Pa and antibiotic-resistant Pa. | over the two-to-five-year observational period
To better define clinical outcomes associated with acquisition of Pa, as well as outcomes associated with emergence of mucoid Pa and antibiotic-resistant Pa. | over the two-to-five-year observational period

SECONDARY OUTCOMES:
Among subjects who acquire Pa but do not enroll in the EPIC Clinical Trial, to examine the effect of the duration of Pa positive respiratory cultures prior to initiation of anti-pseudomonal therapy and the type and length of anti-pseudomonal therapy. | over the two-to-five year observational period
To describe temporal changes in anti-pseudomonal serology and airway microbiology. | over the two-to-five year observational period
To better define clinical outcomes associated with isolation of S. aureus from respiratory cultures, as well as outcomes associated with emergence of methicillin-resistant S. aureus (MRSA). | over the two-to-five year observational period
To bank Pa and S. aureus isolates and serum samples for future studies to enhance the understanding of early CF lung disease. | over the two-to-five year observational period
To use and bank DNA samples for analyses of genetic factors that may be associated with CF pathogenesis, disease progression, and clinical outcomes. | over the two-to-five year observational period
For subjects who enroll in EPIC Clinical Trial, to collect ancillary data on risk factors preceding trial enrollment and to provide follow-up for clinical endpoints after trial participation has ended. | over the two-to-five year observational period
To provide a cohort of subjects who acquire Pa during the observational study period but who do not enroll in EPIC Clinical Trial and therefore receive non protocol-based anti-pseudomonal therapy. | over the two-to-five year observational period

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Rosenfeld, MD, MPH, Principal Investigator — Seattle Children's Hospital; Ronald L. Gibson, MD, PhD, Principal Investigator — Seattle Children's Hospital; Wayne J. Morgan, MD, Principal Investigator — University of Arizona Health Sciences Center
Locations (54):
- United States (54):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Los Angeles / USC Medical School, Los Angeles, California
  - Kaiser Permanente Medical Center, Oakland, California
  - Packard Children's Hosp., Stanford University, Palo Alto, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Denver, Denver, Colorado
  - duPont Hospital for Children, Wilmington, Delaware
  - Nemours Children's Clinic, Jacksonville, Florida
  - All Children's Hospital CF Center, St. Petersburg, Florida
  - Emory University, Cystic Fibrosis Center, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - Riley Hospital, Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Center, Portland, Maine
  - Children's Hospital, Boston, Boston, Massachusetts
  - University of Mass Memorial Health Care, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Spectrum Health Hospitals - DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Hospitals & Clinics, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Hospital - St. Louis University, St Louis, Missouri
  - Washington University School of Medicine/St. Louis Children's Hospital, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Albany Medical College, Albany, New York
  - Women & Children's Hospital of Buffalo, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - University of Rochester, Rochester, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - New York Medical College/Westchester Medical Center, Valhalla, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Rainbow Babies & Childrens Hospital, Cleveland, Ohio
  - Children's Hospital, Columbus, Ohio
  - Children's Medical Center, Dayton, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - LeBonheur Children's Medical Center, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Children's Hospital at Fletcher Allen Health Care, Burlington, Vermont
  - Children's Hospital & Regional Medical Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Rosenfeld M, Emerson J, McNamara S, Thompson V, Ramsey BW, Morgan W, Gibson RL; EPIC Study Group. Risk factors for age at initial Pseudomonas acquisition in the cystic fibrosis epic observational cohort. J Cyst Fibros. 2012 Sep;11(5):446-53. doi: 10.1016/j.jcf.2012.04.003. Epub 2012 May 1. PMID 22554417
- [Derived] Rosenfeld M, Emerson J, McNamara S, Joubran K, Retsch-Bogart G, Graff GR, Gutierrez HH, Kanga JF, Lahiri T, Noyes B, Ramsey B, Ren CL, Schechter M, Morgan W, Gibson RL; EPIC Study Group Participating Clinical Sites. Baseline characteristics and factors associated with nutritional and pulmonary status at enrollment in the cystic fibrosis EPIC observational cohort. Pediatr Pulmonol. 2010 Sep;45(9):934-44. doi: 10.1002/ppul.21279. PMID 20597081
- [Derived] Treggiari MM, Rosenfeld M, Mayer-Hamblett N, Retsch-Bogart G, Gibson RL, Williams J, Emerson J, Kronmal RA, Ramsey BW; EPIC Study Group. Early anti-pseudomonal acquisition in young patients with cystic fibrosis: rationale and design of the EPIC clinical trial and observational study'. Contemp Clin Trials. 2009 May;30(3):256-68. doi: 10.1016/j.cct.2009.01.003. Epub 2009 Jan 15. PMID 19470318